CLINICAL TRIAL: NCT05810090
Title: Functional Outcomes After Total Knee Arthroplasty
Brief Title: The Outcomes of Subject After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 220912
Record Dates: First submitted 2022-10-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-10

CONDITIONS: Satisfaction, Patient
Keywords: Total Knee Arthroplasty (TKA); Western Ontario and McMaster Universities Arthritis Index
MeSH Terms: conditions — Patient Satisfaction | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TKA (Total Knee Arthroplasty): Patients did total knee arthroplasty in our hospital.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — patient who received a TKA in our hospital

SUMMARY:
Total Knee Arthroplasty (TKA) is a standard of intervention for severe knee osteoarthritis, also been proven with benefits in improving pain, mobility, and quality of life. However, the outcomes after TKA is controversial.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) clinical pathway provides preoperative education, postoperative rehabilitation, and routine outpatient follow-up. The overall functional performance of the patient was assessed. The aim of this study was to analyze (1) clinical pain relief, anxiety reduction and functional recovery after TKA; (2) factors affecting individual functional recovery, such as age, gender, BMI, etc.

The results can be used as a reference for improving the quality in TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* unilateral knee TKA

Exclusion Criteria:

* bilateral knee TKA

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data were collected from CCH2000 / TKA clinical pathway databank retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Changes of Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline: date of surgery (day 0); discharge from hospital (D/C), an average of 1 week; 1 month after D/C; 3 months after D/C; 6 months after D/C
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  (I). Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright (II). Stiffness (2 items): after first waking and later in the day (III). Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The assessment was performed at: Baseline: admission date of surgery, discharge from hospital (D/C), 1 month after D/C, 3 months after D/C, 6 months after D/C
Changes of knee Range of motion (ROM) | Baseline: date of surgery (day 0); discharge from hospital (D/C), an average of 1 week; 1 month after D/C; 3 months after D/C; 6 months after D/C
  Range of motion in bilateral Knee joints

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Che Lin, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided